CLINICAL TRIAL: NCT07118488
Title: Multitarget Pulse Field Ablation Guided by Endocardial and Non-invasive Atrial Driver Mapping (PFA+ADM) Pilot Study. Development of an Ablation Strategy to Improve the Efficacy of Long Standing Atrial Fibrillation Ablation in Patients With High Comorbidity Burden or Heart Failure
Acronym: PFA+ADM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Innovacion en Biomedicina (FIBMED) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PFA+ADM
Record Dates: First submitted 2025-07-21; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Persistent Atrial Fibrillation Longstanding
Keywords: Atrial fibrillation; PFA; Rotors; Atrial entanglement; Catheter ablation; ECGi
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm - Multitarget PFA Ablation (Experimental): Pulmonary vein isolation plus extra pulmonary drivers ablation based on EGM findings (rotational and high frequency sites)
  Interventions: Procedure: Multitarget PFA Ablation

INTERVENTIONS:
Procedure: Multitarget PFA Ablation — * Informed consent gave by the patient.
  * Implantable loop recorder procedure
  * Clinical procedure starts
  * Electrophysiologycal study
  * Non-invasive map is obtained.
  * Electroanatomical map of both atria is generated.
  * Intracavitary electrogram (EGM) driver assessment
  * Pulmonary vein isolation
  * Extra pulmonary drivers ablation based on EGM findings (rotational and high frequency sites).
  * Non-invasive map is obtained to assess ablation impact on driver distribution.
  * Remap and extra pulmonary lesions are carried out until activity. At drivers sites disappears or decreases in at least 2 hertz or up to physician criteria.
  * Patient follow up

SUMMARY:
To assess the efficacy and safety of a percutaneous ablation strategy that targets multiple extrapulmonary structures as the Cox-Maze IV.

DETAILED DESCRIPTION:
Persistent and long-standing atrial fibrillation (PsAF and LSAF) remain significant clinical challenges, particularly in patients with heart failure or high comorbidity burden, where the arrhythmia is often more sustained, complex, and resistant to conventional ablation approaches. Despite advancements in ablation technology, pulmonary vein isolation (PVI) alone has shown limited success in this subgroup. Current guidelines acknowledge the need for additional ablation targets beyond the pulmonary veins (PVs), yet evidence remains scarce and optimal strategies undefined.

This single-arm, prospective pilot study investigates a novel ablation strategy that combines multi-target pulsed field ablation (PFA) with both endocardial intracavitary electrogram (EGM) mapping and non-invasive body surface mapping (BSM) to guide the identification and ablation of extra-PV atrial fibrillation drivers. This approach is designed to emulate the multilevel strategy of the surgical Cox-Maze IV, aiming for comprehensive arrhythmia substrate modification while minimizing procedural risk.

The PFA+ADM protocol leverages recent advances in:

* Pulsed Field Ablation (PFA): a non-thermal modality offering selective myocardial ablation with reduced risk to adjacent tissues (e.g., esophagus, phrenic nerve).
* Non-invasive Driver Mapping (ADM): Electrocardiographic imaging (ECGi) with torso vests capable of reconstructing 3D epicardial activation patterns and identifying high-frequency or rotational driver sites.
* Intracardiac Electrogram Analysis: High-resolution EGM signals captured during atrial fibrillation are analyzed to localize driver activity, complex fractionated atrial electrograms (CFAEs), or high dominant frequency regions.

Study Workflow

After informed consent, participants will undergo implantation of an insertable cardiac monitor (ICM) to allow for continuous AF burden tracking. The ablation procedure includes:

1. Baseline Electroanatomical Mapping: Creation of 3D maps of both atria using a high-density mapping catheter.
2. Non-invasive Driver Mapping: Performed using vest-based ECGi systems to non-invasively identify arrhythmogenic sources beyond the PVs.
3. Intracavitary Driver Mapping: Electrograms are analyzed for spectral content, including dominant frequency (DF) and organization index (OI), to confirm rotational or focal drivers.
4. Pulmonary Vein Isolation (PVI): Executed using PFA technology.
5. Targeted Extra-PV Ablation: Ablation of extrapulmonary targets guided by overlap between invasive and non-invasive driver maps. PFA will be used to eliminate identified high-frequency or rotational driver regions.
6. Post-ablation Re-mapping: Repeat non-invasive and invasive mapping to assess residual driver activity and efficacy of lesion sets.
7. Iterative Ablation (if necessary): Further lesion delivery at persistent driver sites, up to a clinically acceptable endpoint, defined as elimination or reduction in dominant frequency by at least 2 Hz or disappearance of driver behavior.
8. Follow-up Assessments: Clinical evaluations and ICM-based rhythm analysis at 3, 6, and 12 months.

Technical Specifics and Rationale

Rationale for Multitarget Approach:

Atrial remodeling in patients with PsAF/LSPsAF is often diffuse and multifocal. Standard PVI addresses the initiating triggers of paroxysmal AF but fails to control perpetuating mechanisms in persistent forms. The multitarget strategy aims to:

* Capture and eliminate active drivers that are not pulmonary in origin.
* Address atrial regions exhibiting consistent high-frequency reentry.
* Improve patient outcomes by personalizing ablation strategy based on individual driver distributions.

Advantages of PFA Technology:

PFA uses irreversible electroporation to ablate cardiomyocytes without significant collateral damage. This is especially relevant when targeting extrapulmonary sites near vulnerable structures (e.g., posterior wall near esophagus, Bachmann's bundle near the aorta). Additionally, PFA has demonstrated faster lesion creation and potentially shorter procedure times with comparable or superior efficacy in preclinical and early clinical data.

Integration of ECGi and EGM-based Mapping:

Simultaneous use of non-invasive ECG imaging and invasive mapping enables comprehensive localization of potential drivers, enhancing ablation precision. The goal is to improve arrhythmia control without significantly increasing procedural complexity or risk.

Patient Profile and Unmet Needs:

This trial targets patients often excluded or underrepresented in clinical trials-those with heart failure or multiple comorbidities who have higher recurrence rates post-ablation. These patients also tend to have more advanced atrial myopathy and may benefit from a more aggressive substrate modification strategy, if delivered safely.

Data Handling and Interim Analysis

Data will be collected prospectively, including electrogram recordings, ECGi maps, procedural data, imaging, and follow-up rhythm status. An interim analysis is planned after the first 25 patients to evaluate safety and refine the mapping-ablation workflow if necessary. Data from ICMs will be analyzed to calculate daily AF burden, detect arrhythmia recurrence, and correlate clinical outcomes with procedural findings.

Safety is evaluated both acutely and in follow-up, with predefined thresholds for major complications (≤5%). The use of PFA is expected to significantly reduce thermal injury risks. Procedural metrics such as total duration, fluoroscopy time, and energy delivery time will also be recorded.

This pilot study will serve as a foundation for larger multicenter trials by assessing the feasibility and clinical benefit of this precision-guided, multitarget ablation strategy in a high-risk AF population. Its results may help redefine ablation endpoints beyond pulmonary vein isolation and facilitate the integration of novel technologies into routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80.
* Ability and willingness to follow the study protocol, including informed consent.
* Symptomatic long-standing AF for at least one month, documented by ECG or dual-chamber device recordings.
* History of failure, intolerance, or refusal of antiarrhythmic drug therapy.
* New York Heart Association (NYHA) functional class II or III, or left ventricular dysfunction (LVEF ≤ 50%) or a CHA2DS2-VASc score of 4 or more.
* Optimal medical treatment for heart failure for at least three months for patients with left ventricular dysfunction.

Exclusion Criteria:

* Left atrial diameter >5.5 cm.
* Previous left atrial ablation or surgery.
* Lack of anticoagulation therapy for 3 weeks prior to the procedure.
* Pulmonary vein stents or stenosis.
* Pre-existing diaphragmatic paralysis.
* Cardiac valve prosthesis or significant valve disease.
* Recent cardiac surgery or interventions within the past 3 months.
* Unstable angina, NYHA Class IV heart failure.
* Pulmonary hypertension or rheumatic heart disease.
* Blood clotting disorders.
* Contraindications to chronic anticoagulation.
* Active infection or hypertrophic cardiomyopathy.
* Reversible causes of AF, such as hyperthyroidism or sleep apnea.
* Stroke or TIA in the past 6 months.
* History of thromboembolic events or evidence of intracardiac thrombus.
* Women of childbearing age
* Life expectancy less than 12 months.
* Participation in another clinical trial.
* Allergy to adhesives.
* Inability to comply with study procedures.
* Inability to provide personal consent.
* NYHA Class IV heart failure.
* Left ventricular ejection fraction ≤ 25%.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of Successful Pulmonary Vein Isolation and Freedom from Atrial Fibrillation or Reduction in Arrhythmia Burden | 1 year
  Success is defined as complete isolation of all pulmonary veins and either absence of atrial fibrillation recurrence or a significant reduction in arrhythmia burden over a 1-year follow-up period.
Incidence of Procedure-Related Complications, Including Mortality, Pulmonary Vein Stenosis, Nerve Injury, Stroke, and Major Bleeding Events [Safety] | 6 months
  The safety endpoint is defined as maintaining a complication rate of ≤5%, assessed by monitoring for acute and long-term complications such as mortality, pulmonary vein stenosis, nerve injury, stroke, bleeding, and other serious adverse events occurring within 30 days to 6 months post-procedure.

SECONDARY OUTCOMES:
Percentage of patients in Per AF at the end of follow-up | 1 year
  Percentage of patients in Per AF at the end of follow-up.
Time to the first episode of atrial arrhythmia of more than 30 seconds | 1 year
  Time to the first episode of atrial arrhythmia of more than 30 seconds
Percentage of patients with AF/AT recurrence | 1 year
  Percentage of patients with AF/AT recurrence
Percentage of patients with <50% of AF/AT burden | 1 year
  Percentage of patients with <50% of AF/AT burden
Left ventricular end-systolic volume at the end of follow-up | 1 year
  Physician assessment to measure the function parameters and ventricular size at the end of follow-up using ECHO or MRI. Left ventricular end-systolic volume at the end of 12-month follow-up. Units in mL.
Left ventricular end-diastolic volume at the end of follow-up | 1 year
  Physician assessment to measure the function parameters and ventricular size at the end of follow-up using ECHO or MRI. Left ventricular end-diastolic volume at the end of 12-month follow-up. Units in mL.
Left ventricular ejection fraction (LVEF) at the end of follow-up | 1 year
  Physician assessment to measure the function parameters and ventricular size at the end of follow-up using ECHO or MRI. Left ventricular ejection fraction (LVEF) at the end of 12-month follow-up. Units in percentage.
NYHA Functional Class at the end of follow-up | 1 year
  NYHA Functional Class at the end of follow-up
Adverse events of the procedures | 1 year
  Death, peripheral embolism, stroke, and plugging
Procedure duration/fluoroscopy time | Measured on the day of the ablation procedure. No time frame.
  Procedure duration/fluoroscopy time
Unplanned hospital admission for cardiovascular reasons | 1 year
  Unplanned hospital admission for cardiovascular reasons during the 12-month follow-up after the ablation procedure.
Unplanned hospital admission for any reason | 1 year
  Unplanned hospital admission for any reason during the 12-month follow-up after the ablation procedure.
New onset heart failure | 1 year
  New onset heart failure during the 12-month follow-up after the ablation procedure.
Worsening of functional class due to heart failure | 1 year
  Worsening of functional class due to heart failure during the 12-month follow-up after the ablation procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Angel Arenal, MD, PhD, Principal Investigator — Hospital General Universitario Gregorio Marañón
Locations (1):
- Hospital General Universitario Gregorio Marañon, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No